CLINICAL TRIAL: NCT00792363
Title: A Phase II Study of Irinotecan and Panitumumab as 3rd Line Treatment of Patients With Metastatic Colorectal Cancer Without KRAS Mutations
Brief Title: Irinotecan and Panitumumab as 3rd Line Treatment for mCRC Without KRAS Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2008-004923-48; S-20080104; DKMA 2612-3844
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: KRAS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Irinotecan — 350 mg/m2 intravenously on day 1 every 3 weeks
Drug: Panitumumab — 9 mg/kg intravenously on day 1 every 3 weeks

SUMMARY:
The purpose of this study is to investigate the effect and the side effect profile of irinotecan and panitumumab administered every 3 weeks as 3rd line treatment for patients with metastatic colorectal cancer without KRAS mutations.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most frequent types of cancer in Denmark with approximately 3,400 diagnosed patients per year. The prognosis for these patients is still very poor and more than half of them will develop metastatic disease and thus be candidates for chemotherapy.

In Denmark 5-FU and Oxaliplatin or Irinotecan has been used for several years either as combination or mono therapy. In recent years biological antibodies targeted against EGFR have been added to this treatment. A newly developed antibody is Panitumumab, which enables treatment every 3 weeks instead of weekly administration.

The effect of EGFR activation is mediated through intracellular pathways involving the KRAS protein. It has been proven that a mutation of KRAS causes the KRAS protein to be constantly activated, and patients with these mutations do not benefit from antibodies against EGFR. Approximately 40% of the patients present these mutations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma in colon or rectum with metastatic spread.
* No mutations in the KRAS gene.
* Resistance to 5-FU, oxaliplatin and irinotecan.
* Age ≥18 years.
* PS 0-2.
* Measurable disease according to RECIST criteria.
* Haematology: Neutrophilocytes ≥1.5 x 109/l, leukocytes ≥3.0 x 109/l, thrombocytes ≥100 and bilirubinaemia ≤3 x upper normal value. Samples no more than 4 weeks old.
* Fertile women must present a negative pregnancy test and use secure birth control during and 3 months after treatment.
* Acceptance that blod and tissue samples are kept for subsequent investigation of biomarkers.
* Oral and written informed consent.

Exclusion Criteria:

* Other malignant disease within the past 5 years, excl. non-melanoma skin cancer and carcinoma in situ cervicis uteri.
* Chemotherapy, radiotherapy or immunotherapy within the past 4 weeks.
* Verified or clinically suspected CNS metastasis.
* Other experimental treatment.
* Serious medical disease according to investigator's judgement.
* Pregnant or breastfeeding women.
* Hypersensitivity to the active substance or to one or more of the auxiliary substances.
* Patients with interstitial pneumonitis or pulmonary fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Response Rate | Every 9 weeks. Up to 6 months

SECONDARY OUTCOMES:
Overall survival | 6 months
Progression free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, Professor, Study Chair — Vejle Hospital
Locations (1):
- Vejle Hospital, Dept. of Oncology, Vejle, Denmark